CLINICAL TRIAL: NCT03901872
Title: Contemporary Endovascular Therapies in Treatment of Acute Iliofemoral Deep Vein Thrombosis A Prospective, Multicentre Cohort Trial A Physician Initiated Research Study Request
Brief Title: Contemporary Endovascular Therapies in Treatment of Acute Iliofemoral Deep Vein Thrombosis
Acronym: CLEAR-DVT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS 254427
Record Dates: First submitted 2019-04-02; First posted 2019-04-03 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-04

CONDITIONS: Thrombolysis; Deep Vein Thrombosis
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Acute Iliofemoral DVT: Suitable patients would be invited to take part in this trial as part of standard of care.
  Interventions: Device: Contemporary endovascular venous intervention by Zelante pharmacomechanical thrombolysis

INTERVENTIONS:
Device: Contemporary endovascular venous intervention by Zelante pharmacomechanical thrombolysis — All patients will undergo ultrasound guided micro puncture venous access of the enrolled ipsilateral lower extremity popliteal vein followed by a diagnostic venogram to define thrombus burden and anatomic extent of DVT. Prior to and every 30 minutes during the endovascular procedure, an activated clotting time (ACT) will be obtained. Intravenous unfractionated heparin will be administered to keep the ACT between 250 - 300. A Zelante catheter will be utilised to perform pharmacomechanical thrombolysis of the enrolled lower extremity. If there is involvement of the popliteal and/or femoral vein, pharmacomechanical thrombolysis should also be performed of these veins. Venous stenting may be implemented to address areas of residual venous stenosis or outflow obstruction following pharmacomechanical thrombolysis. Stent placement in the common iliac, external iliac, and common femoral vein are routinely done to address inflow or outflow issues after pharmacomechanical thrombolysis.

SUMMARY:
The goal of this initial proof of principle single arm cohort trial is to determine if contemporary endovascular venous intervention, compared with a 1:1 propensity-matched medical therapy arm of the ATTRACT trial, significantly reduces the 2-year occurrence of Post Thrombotic Syndrome (PTS) in subjects with symptomatic proximal Deep Vein Thrombosis (DVT).

DETAILED DESCRIPTION:
A single arm cohort will serve as a proof of principle study, and be the foundation for a larger subsequent prospective, Randomised Clinical Trial (RCT). The aim of this initial single arm cohort is to both validate that contemporary catheter directed therapy performed by experienced operators has significant efficacy and safety at 10 days, 30 days, 6 months, 12 months, and 2 years (details below). If a strong signal of efficacy and safety is found in the initial single arm cohort at 30 days and 6 months, this will provide objective evidence to move forward with a larger multicentre, prospective, RCT.

If the results of the initial single arm proof of principle cohort do not show efficacy, or there is a safety issue, a larger prospective, RCT will not be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patient age 16 years to 75 years.
* Onset of acute DVT symptoms of 14 days or less in the study limb.
* DVT located in the common and/or external iliac, or common femoral vein
* Consent to participate in this research study and be willing to commit to study requirements including completion of questionnaires and follow-up visits.

Exclusion Criteria:

* In the index leg: established PTS, or previous symptomatic DVT within the last 2 years.
* In the contralateral (non-index) leg: symptomatic acute DVT a) involving the iliac and/or common femoral vein; or b) for which thrombolysis is planned as part of initial therapy.
* Limb-threatening circulatory compromise.
* Pulmonary embolism defined as either massive (Systolic blood pressure < 90 mmHg and/or patient on IV vasoactive medication to support blood pressure), or intermediate high risk pulmonary embolism (PE), as defined by the European Society Guideline on management of PE. Low risk PE and/or intermediate low risk PE can be enrolled.
* Inability to tolerate contemporary venous intervention procedure due to severe dyspnea or acute systemic illness.
* Allergy, hypersensitivity, or thrombocytopenia from heparin, Recombinant tissue plasminogen activator (rtPA), or iodinated contrast, except for mild-moderate contrast allergies for which steroid pre-medication can be used.
* Haemoglobin < 9.0 mg/dl, INR > 1.6 before starting anticoagulation, or platelets < 100,000/ml. Moderate renal impairment in diabetic patients (estimated glomerular filtration rate < 60 ml/min) or severe renal impairment in non-diabetic patients (estimated glomerular filtration rate < 30 ml/min).
* Active bleeding, recent (< 3 mo) GI bleeding, severe liver dysfunction, bleeding diathesis.
* Recent (< 3 mo) internal eye surgery or haemorrhagic retinopathy; recent (< 10 days) major surgery, cataract surgery, trauma, cardiopulmonary resuscitation, obstetrical delivery, or other invasive procedure.
* History of stroke or intracranial/intraspinal bleed, tumor, vascular malformation, aneurysm.
* Active cancer (metastatic, progressive, or treated within the last 6 months). Exception: patients with non-melanoma primary skin cancers are eligible to participate in the study.
* Severe hypertension on repeated readings (systolic blood pressure > 180 mmHg or diastolic blood pressure > 105 mmHg). This can be treated, and blood pressure must be stable before venous access is obtained (systolic blood pressure <140 mmHg).
* Pregnant (positive pregnancy test, women of childbearing potential must be tested).
* Recently (< 1 mo) had thrombolysis or is participating in another investigational device or drug study that may convolute study results.
* Life expectancy < 2 years or chronic non-ambulatory status.
* Inability to provide informed consent or to comply with study assessments (e.g. due to cognitive impairment or geographic distance).
* Inferior vena cava (IVC) thrombus. Significant thrombus of the IVC, by definition, thrombus extending more than one centimeter above the IVC - common iliac vein confluence will be a cause for exclusion.
* Inability to obtain access of the enrolled ipsilateral popliteal vein using ultrasound guided micro-puncture technique.
* History of, or active heparin induced thrombocytopenia (HIT).

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All acute DVT patients will be screened for entry into the trial
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2019-03-29 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Rate of Post thrombotic Syndrome at 2 years | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Guy's & St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided